CLINICAL TRIAL: NCT04668534
Title: Effect of Transcutaneous Auricular Vagal Nerve Stimulation on Functional Dyspepsia: a Randomized Controlled Trial
Brief Title: Effect of Transcutaneous Auricular Vagal Nerve Stimulation on Functional Dyspepsia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Yanglin Pan, Associated professor, Air Force Military Medical University, China
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KY20202087-F-1
Record Dates: First submitted 2020-12-06; First posted 2020-12-16 (Actual); Last update posted 2020-12-16 (Actual); Status verified 2020-12

CONDITIONS: Functional Dyspepsia
Keywords: Functional Dyspepsia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment group 1 (Experimental): Based on the infection of Hp or not, patients will receive quadruple therapy (amoxicillin, clarithromycin, pantoprazole, and bismuth) or PPI (pantoprazole) plus taVNS (produced by by Xi'an Bashui Health Technology Co., Ltd) at left tragus. Patients were given taVNS thirty minutes twice a day in the morning and the night for four weeks (duty circle: 30s "on" periods and 30s "off" periods; frequency: 10 Hz; current intensity: minimal pain threshold; pulse width: 500 μs).
  Interventions: Device: taVNS 10
- Treatment group 2 (Experimental): Based on the infection of Hp or not, patients will receive quadruple therapy (amoxicillin, clarithromycin, pantoprazole, and bismuth) or PPI (pantoprazole) plus taVNS (produced by by Xi'an Bashui Health Technology Co., Ltd) at left tragus. Patients were given taVNS thirty minutes twice a day in the morning and the night for four weeks (duty circle: 30s "on" periods and 30s "off" periods; frequency: 25 Hz; current intensity: minimal pain threshold; pulse width: 500 μs).
  Interventions: Device: taVNS 25
- Control group (Active Comparator): Based on the infection of Hp or not, patients will receive quadruple therapy (amoxicillin, clarithromycin, pantoprazole, and bismuth) or PPI (pantoprazole) plus taVNS (produced by by Xi'an Bashui Health Technology Co., Ltd) at left earlobe. Patients were given taVNS thirty minutes twice a day in the morning and the night for four weeks (duty circle: 30s "on" periods and 30s "off" periods; frequency: 10 Hz; current intensity: minimal pain threshold; pulse width: 500 μs).
  Interventions: Device: Control

INTERVENTIONS:
Device: taVNS 10 — Patients were given taVNS (by Xi'an Bashui Health Technology Co., Ltd) thirty minutes twice a day in the morning and the night for four weeks (duty circle: 30s "on" periods and 30s "off" periods; frequency: 10 Hz; current intensity: minimal pain threshold; pulse width: 500 μs)
  Arms: Treatment group 1
Device: taVNS 25 — Patients were given taVNS (by Xi'an Bashui Health Technology Co., Ltd) thirty minutes twice a day in the morning and the night for four weeks (duty circle: 30s "on" periods and 30s "off" periods; frequency: 25 Hz; current intensity: minimal pain threshold; pulse width: 500 μs)
  Arms: Treatment group 2
Device: Control — Patients were given taVNS (by Xi'an Bashui Health Technology Co., Ltd) thirty minutes twice a day in the morning and the night for four weeks (duty circle: 30s "on" periods and 30s "off" periods; frequency: 10 Hz; current intensity: minimal pain threshold; pulse width: 500 μs)
  Arms: Control group

SUMMARY:
Patients with dyspeptic symptoms vary from 10% to 20% globally. Up to 70% of patients with dyspepsia who undergo endoscopy have unremarkable examination and are diagnosed with functional dyspepsia (FD). Given the lack of information related to its pathophysiology, the treatment is largely empirical and of limited efficacy. Previous small study showed therapeutic potential of transcutaneous auricular vagal nerve stimulation (taVNS) for FD. This study aims to investigate whether taVNS can improve the dyspeptic symptoms of patients with FD.

ELIGIBILITY:
Inclusion Criteria:

1. 18-65 years old
2. Patients who met the Rome IV diagnostic criteria of FD
3. Moderate to severe FD (functional dyspepsia symptom diary ≥10)
4. Normal upper endoscopy and abdominal ultrasonography within one year.

Exclusion Criteria:

1. Injury or inflammation on the ear
2. Asthma or COPD not under control
3. History of cardiac pacemaker planting or other medical digital devices
4. History of VNS treatment
5. Patients with local or systemic diseases which may cause dyspeptic symptoms:

   Known active peptic ulcer, cholecystitis, gallstone, gastrointestinal obstruction, gastroparesis, and etc.; Known acute or chronic injury of liver or kidney; Obvious hematological abnormality, or endocrine and metabolic diseases; Known malignancy; Obvious cardiovascular or cerebrovascular diseases (such as coronary heart disease, arrhythmia, cerebral infarction and etc.; Other conditions which may be associated with dyspeptic symptoms (such as NSAIDs associated dyspepsia)
6. Patients with serious mental disorders or tendency to suicide
7. Pregnancy or lactic women
8. Inability to give informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-12-28 (Estimated); Study Completion 2022-03-28 (Estimated)

PRIMARY OUTCOMES:
Responder rate | 4 weeks
  The proportion of patients whose Functional Dyspepsia Symptom Diary Total Symptom Scores were reduced ≥5 after four weeks treatment when compared with baseline.

SECONDARY OUTCOMES:
Functional Dyspepsia Symptom Diary (FDSD) | 4 weeks
  The FDSD consists of 5 cardinal items (burning in the stomach, stomach pain, bloating, postprandial fullness, and early satiety) and 3 supplementary items (nausea, burping/belching rating, and burping/belching bother). Each item can be scored from 0 (no) to 10 (worst). Total Symptom Score includes the 5 cardinal items and ranges from 0 to 50.
Gastrointestinal Symptom Rating Scale (GSRS) | 4 weeks
  The GSRS contains 15 items. All individual items are scored on a 7-point Likert scale (1 = not at all to 7 = extremely) and are subsequently clustered into five domains (abdominal pain, reflux, indigestion, diarrhea, and constipation); higher scores indicate more severe symptoms.
Adequate relief rate | 4 weeks
  The proportion of patients who acquire overall symptom relief when compared with baseline
Elimination rate of cardinal symptom | 4 weeks
  The proportion of patients whose cardinal symptom is completely eliminated when compared with baseline.

OTHER OUTCOMES:
Short Form of Nepean Dyspepsia Index (SF-NDI) | 4 weeks
  The SF-NDI consists of 10 questions regarding the effects of dyspepsia symptoms ("stomach problems") on different aspects of life (tension, interference with daily activities, eating/drinking, knowledge/control, and work/study). Each response can be from 1 (not at all affected) to 5 (extremely affected), or 0 (N/A), for a total summed score out of 50.
Hamilton Anxiety and Depression Scale | 4 weeks
  Anxiety and depression of patients are assessed by using Hamilton Anxiety and Depression Scale.
  Hamilton Anxiety Scale consists of 14 items. Each item is scored on a scale from 0 (absent) to 4 (most severe) with a total score range of 0-56.
  Hamilton Depression Scale consists of 17 items. Individual items scored on 3 point (0 to 2) or 5 point scale (0 to 4); 0=absent, 4=most severe. Total score: 0 to 52.
Adverse event | 4 weeks

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Lanzhou University Second Hospital, Lanzhou, Gansu
  - Xijing Hospital of Digestive Diseases, Xi'an, Shaanxi
  - The Second Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi

IPD SHARING:
Plan to Share IPD: No
Other researchers can contact PI to get IPD.

REFERENCES:
- [Derived] Shi X, Zhao L, Luo H, Deng H, Wang X, Ren G, Zhang L, Tao Q, Liang S, Liu N, Huang X, Zhang X, Yang X, Sun J, Qin W, Kang X, Han Y, Pan Y, Fan D. Transcutaneous Auricular Vagal Nerve Stimulation Is Effective for the Treatment of Functional Dyspepsia: A Multicenter, Randomized Controlled Study. Am J Gastroenterol. 2024 Mar 1;119(3):521-531. doi: 10.14309/ajg.0000000000002548. Epub 2023 Oct 3. PMID 37787432